**PRINCIPAL INVESTIGATOR:** Christine Alewine, M.D., Ph.D.

STUDY TITLE: A Phase II Trial of the Superenhancer Inhibitor Minnelide

in Advanced Refractory Adenosquamous Carcinoma of

the Pancreas (ASCP)

STUDY SITE: NIH Clinical Center

Cohort: *Affected patient – Standard* 

Consent Version: 06/27/2023

## WHO DO YOU CONTACT ABOUT THIS STUDY?

**Principal Investigator:** Christine Alewine, M.D., Ph.D.

#### KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you in making your decision about participating in this study. Additional information that may help you decide can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to take part in this study because you have adenosquamous carcinoma of the pancreas (ASCP) or high suspicion for ASCP.

The purpose of this consent form is to describe how treatment on the clinical trial will happen. You have completed screening and were found to be eligible for treatment on the study, if you choose to do so. The purpose of this treatment part of the study is see if using Minnelide may be a better way to treat your cancer.

The use of Minnelide in this study is considered investigational, which means that it has not been approved by the U.S. Food and Drug Administration (FDA) to treat ASCP. However, the FDA has given us permission to use Minnelide in this study.

There may be other drugs that may be used to treat your disease, and these can be prescribed/given by your regular cancer doctor, even if you are not in this study. The way in which treatment is given in this study and the side effects are not significantly different than if you were to receive standard care therapy.

If you decide to join this study, here are some of the most important things that you should know that will happen:

We will first do some basic tests to make sure you still qualify for the trial.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Version Date:06/27/2023




- You will take Minnelide by mouth every day for 21 consecutive days each cycle. Each cycle of treatment is 28 days and there will be a 7-day resting period between cycles. Treatment may continue for a total of 12 cycles.
- You may experience side effects from taking part in this study. Some can be mild or very serious, temporary, long-lasting, or permanent, and may include death. Examples of some of the side effects that you may have include low blood counts which could affect your ability to fight infection, fatigue and nausea. Other side effects are described further on in this consent form. It is important that you read these
- You will be seen regularly during the study. You will have clinical, laboratory, and imaging tests to see how you are doing and to assess your disease. We will also collect required samples from you (such as blood and tissue) for both clinical and research purposes.
- After the study treatment has ended, we will ask you to come to the NIH Clinical Center for a follow-up visit. If this is not possible, we will contact you or your physician by telephone to collect clinical data and ask about any other cancer therapies you may have started and about your survival status.
- If you are capable of becoming pregnant or you are a sexually active person with a partner capable of becoming pregnant, you and your partner must agree to use birth control before initiating the study, during the study. If you are female, you must continue this birth control for 6 months after the last dose of treatment. If you are male, you must continue this birth control for 3 months after the last dose of treatment.

Just as we do not know what side effects you might have, we cannot know if you may benefit from taking part in this study. If you do not benefit, this study and the results from our research will help others in the future.

You are free to stop participating in the trial at any time. If you decide to stop, the study doctor may ask you to agree to certain tests to make sure it is safe for you to stop.

The remaining document will now describe the research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about the information in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research interventions in which they would want to participate. Take the time you need to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

# IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17) File in Section 4: Protocol Consent (2) Version Date:06/27/2023 



#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to see if Minnelide is an effective treatment for ASCP.

We are asking you to join this research study because you have been diagnosed with ASCP or high suspicion for ASCP and your cancer did not respond to previous therapies.

Minnelide is considered investigational, which means that it has not been approved by the U.S. Food and Drug Administration (FDA) to treat ASCP. We are testing it in this research study to see if it could be used to treat your cancer.

#### WHAT WILL HAPPEN DURING THE STUDY?

The screening process showed that you are eligible to participate in the study, and if you choose to be in it, you may need to have a few additional standard tests completed if not done recently. You will also have additional samples collected for research tests. If any of the screening tests need to be repeated, and show that you have become ineligible, you will not be able to continue with this study.

If you decide to take part in the study, you will be asked to:

- Receive study treatment at the NIH Clinical Center and be seen regularly in the clinic, to have tests and procedures during and after the study treatment in follow-up to see how you are doing and to assess your disease
- Provide specimens (such as blood, tumor and normal tissue) for research studies.

# **Study Treatment**

The study is divided up into segments of time called "cycles". For this study, a cycle will be 28 days.

Minnelide will be taken once daily for 21 consecutive days for each cycle. Each cycle of treatment is 28 days and there will a 7 day resting period between cycles. The capsules must be stored in the refrigerator. The capsule must be swallowed whole with one cup of water and should not be chewed. You should take Minnelide at approximately the same time every day and you should not eat for at least 30 minutes prior and 90 minutes after Minnelide administration. If you forget to take Minnelide, you will not take the missed dose if it is more than 6 hours late.

Before you start taking any new medicines, including medicines you can buy 'over-the-counter', please talk to the study doctor to make sure they are allowed on this study. You will be asked to keep a diary of the medicine that you are taking during the study. We will be reviewing this diary with you during your visits to the clinic, so please bring it to every visit.

At each clinic visit at the NIH Clinical Center, please bring your completed medication diary pages and all of your capsule containers (whether they are empty or not) as we will be counting the capsules and reviewing your diary pages as part of the safety evaluation for this study.

If you have certain side effects, the dose of Minnelide may be held or reduced to prevent return of the side effect. If the side effect(s) is/are too severe, Minnelide may need to be stopped.

You may continue receiving Minnelide for a maximum of 12 cycles or as long as your disease does not get worse and you do not have serious side effects or you decide to stop receiving the study treatment.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




While you are taking study medication, we will perform some tests and examinations for safety and to test the effect of the study therapy. You will need to be seen in clinic at the NIH Clinical Center about every 2 weeks for the first cycle, then at least at the beginning of each cycle after. We will check on you by phone to see how you are doing on the other weeks in the first cycle, then in the middle of each cycle after. If needed, you may be asked to come to clinic more often. At every visit (phone or in-person) you will get labs at the NIH or closer to home. See additional testing below. We will also collect samples from you for purposes of research only. The assessments and tests to be done include:

- Physical exams and measures of your vital signs. You will also be asked about any changes in medications that you are taking and changes in how you are feeling to check for potential side effects.
- Performance status
- Pregnancy test if you are able to become pregnant. Lab blood (up to 1 tablespoon/visit) and urine tests
- Blood for tumor markers (about ½ tablespoon)
- Imaging with CT and/or MRI will be done to assess the sites of your disease at the beginning of every other cycle.

## Additional research testing

In addition to the tests that we will conduct to determine whether you are having side effects or if you are responding to the study therapy, we will also collect samples from you for purposes of research only. The samples are being done to look at the effects of therapy on markers of tumor activity.

The samples included for these studies include:

- Blood
- Required tumor tissue collected before you start treatment this may be tissue from a prior biopsy or procedure within the last 90 days, after any prior treatment. If this tissue is not available, you will be required to have a biopsy for the study prior to treatment.
- Optional tumor biopsy collected before you start treatment (required if tissue is not available from a prior procedure), during cycle 1 and at the end of treatment.

All of your samples collected for research purposes on this study (such as the tumor and normal tissue) may be used to look for specific changes in the DNA in tumors that could be used to develop new ways of diagnosing and treating cancer. DNA (also called deoxyribonucleic acid) in the cells carries genetic information and passes it from one generation of cells to the next - like an instruction manual. Normal tissue contains the DNA (instructions) that you were born with, DNA in tumor cells has changed – or mutated – and we think that change in the DNA is what causes tumors to form and to grow.

To look at your DNA, we may use what is called "whole genome sequencing." This is where we will do special tests in the lab to look at the entire sequence, or order, of how your DNA is put together. This is what makes you unique.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




To determine which parts of the DNA have mutated, we will compare the DNA in your tumor cells to DNA from your normal cells. We will then analyze the results from similar tumors to see if there are any changes in the DNA that are common to a particular type of tumor. To examine the tumor and normal tissue we may use several different techniques depending on the type of tissue we collect. These could include growing cell lines (cells which keep dividing and growing in the laboratory, sometimes for years allowing us to continually study those cells), xenograft studies (placing or growing cells in another animal, such as mice), and looking in detail at the parts of the genes that produce specific proteins.

However, you should know that the analyses that we perform in our laboratory are for research purposes only; they are not nearly as sensitive as the tests that are performed in a laboratory that is certified to perform genetic testing or testing for routine clinical care. For these reasons, we will not give you the results of the research tests done on your research samples in most cases. There may be exceptions to what we share with you and this is described later in this consent form in the section for "Return of research results."

# When you are finished taking the drugs

If you need to stop participating in the study treatment for any reason (including that your disease has started to grow while you are receiving the treatment), then you will be asked to return to the NIH no later than about 4 weeks after you have had last dose of study drug and before you begin a new anti-cancer treatment for an end of treatment visit.

The visit will include the following clinical tests:

- Physical exam including weight and vital signs
- Performance status
- Electrocardiogram
- Lab blood and urine tests
- Pregnancy test if you are a woman who can have children
- CT Scans and/or MRI (if not within the last 4 weeks).
- Blood for tumor markers

If you are unable to return to NIH for this visit, we may contact you or your local physician to collect clinical data and ask for your symptoms.

## HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this study, your involvement is expected to last for one year or until your cancer worsens, you have unacceptable side effects, you decide to no longer take part in the study, or your study doctor decides it is no longer suitable for you to continue.

You will be seen several times during treatment. The outpatient visits during and after treatment usually take about 3 hours but should not take longer than 8 hours.

#### HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

We plan to have approximately 55 people participate in this study at the NIH.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




#### WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

If you choose to take part in this study, you are at risk for side effects. The study doctors do not know who will or will not have side effects. Some side effects may go away soon, some may last a long time, and some may never go away. It is also possible that you may experience more than one side effect at the same time. Some side effects may be mild. Other side effects may be very serious and even result in death.

Minnelide should not be taken together with certain medications, such as those often taken for nausea and vomiting. Please note that Minnelide should not be taken with medications that contain ondansetron (also known as Zofran). Be sure to talk with your doctor or another member of the study team prior to taking ondansetron or any other new medications.

#### Risks and Possible Side Effects of Minnelide

- Reduction of numbers of blood cells potentially resulting in:
  - o Decreased ability of the immune system to fight infection which could lead to hospitalization for serious, life-threatening infection or death. Fatal infection has been observed following treatment with Minnelide
  - Decreased ability to clot blood
  - o Anemia (decrease in the number of red blood cells)
- Changes in your digestion or activity of your stomach and/ or bowels causing:
  - o Abdominal pain, nausea, or vomiting
  - Diarrhea or constipation
  - Weight loss
  - o Dehydration
  - Decreased appetite
  - **Tiredness**

If you experience a combination of these side effects at the same time, you may need extra fluids to protect your kidneys. Call your study team immediately if this occurs.

Decreases in the concentrations of sodium, potassium or phosphate in your blood which may require supplementation by pill or infusion.

Rare but serious

Changes in speech, balance, gait, swallowing and limb coordination

#### **Risks from Study Research Procedures**

The following study procedures and treatments may have risks and cause discomfort while you participate on this study:

#### **Blood draws**

Risks include temporary discomfort, pain, redness, bleeding, bruising, and swelling at the site where the needle is inserted, and/or very rarely inflammation/infection of the vein, which could require antibiotics. You may also experience dizziness, nausea, or rarely, fainting during blood taking. Please tell the study doctor if you do not feel well after having your blood drawn. We will

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




not collect more than 4 tablespoons of blood during any day of study or 12 tablespoons within 8 weeks.

#### Urine collection

There is no risk related to urine collection.

# Electrocardiogram (ECG)

Some skin irritation can occur where the ECG/EKG electrodes are placed. Once the electrodes are placed, the test will begin, is completely painless, and generally takes less than a minute to perform. After the test, the electrodes are removed.

## **Tumor biopsies (optional)**

If your doctor determines it is safe we may obtain a piece of your tumor (biopsy) using a needle with minimal risk to you. You will be given local anesthesia (numbing medicine) and a sedative prior to the biopsy. The biopsy will be taken through a needle put through the skin into your tumor. Depending upon the location of your tumor, a CT scan may be used to assist the biopsy. After the procedure the nurses will watch your blood pressure and other vital signs.

There may be some temporary pain or discomfort during the procedure and afterwards in the area where the tissue was removed. You may also experience some bruising around the biopsy site over the following days. In rare cases an infection or bleeding may occur.

## **Imaging**

In addition to the radiation risks discussed below, CT scans may include the risks of an allergic reaction to the contrast. Participants might experience hives, itching, headache, difficulty breathing, increased heartrate and swelling.

#### Risks for MRI

Magnetic resonance imaging (MRI) uses a strong magnetic field and radio waves to take pictures of the body. We will obtain pictures of your chest, abdomen and pelvis for this study. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




IRB APPROVAL DATE: 6/27/2023

having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

#### Risks from Gadolinium

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (IV) catheter (small tube). It will be done for both research and medical purposes.

It is not known if MRI with contrast is completely safe for a developing fetus. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each MRI scan with contrast. The scan will not be done if the pregnancy test is positive.

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis (NSF)". This condition always involves the skin and can also involve the muscles, joints and internal organs. NSF has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is below the safe level.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA has issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain in the body than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain in the body.

## What are the risks related to pregnancy?

If you are able to become pregnant, we will ask you to have a pregnancy test before starting this study. You must use effective form of birth control methods and try not to become pregnant during study treatment, and for 6 months after you finish study treatment. If you become pregnant, there may be unknown risks to the fetus or unborn child, or risks that we did not anticipate. There may be long-term effects of the treatment being studied that could increase the risk of harm to a fetus. You must tell the study doctor if your birth control method fails during the restricted period. If you think or know you have become pregnant while participating in this research study, please contact the study team as soon as possible. If you plan to become pregnant in the future, please discuss

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




with the study team how long you need to wait before becoming pregnant after completing the study.

If you are a sexually active person with a partner able to become pregnant, it is important that your partner not become pregnant during study treatment, and for 3 months after you finish study treatment. There may be unknown risks to a fetus or risks we did not anticipate. You and your partner must agree to use birth control if you want to take part in this study. If you think your partner has become pregnant during the restricted period, please contact the study team as soon as possible. If you and your partner plan for your partner to become pregnant after your participation in this study, please discuss this with the study team.

# What are the risks of radiation from being in the study?

During your participation in this research study, you may be exposed to radiation from up to 3 CT guided biopsies, and up to 4 CT scans. The amount of radiation exposure from these procedures is equal to approximately 7.6 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The CT guided biopsies and CT scans that you get in this study will expose you to the roughly the same amount of radiation as 25.3 years' worth of background radiation. Being exposed to too much radiation can cause harmful side effects such as an increase in the risk of cancer. The risk depends on how much radiation you are exposed to. Please be aware that about 40 out of 100 people (40%) will get cancer during their lifetime, and 20 out of 100 (20%) will die from cancer. The risk of getting cancer from the radiation exposure in this study is 0.8 out of 100 (0.8%) and of getting a fatal cancer is 0.4 out of 100 (0.4%).

You may not participate in this study if you are pregnant. If you are able to become pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

#### **Privacy Risks Associated with Genetic Testing**

It may be possible that genetic information from you could be used by law enforcement agencies or other entities to identify you or your blood relatives

# Psychological or Social Risks Associated with Return of Incidental or Secondary Findings

As part of the research study, it is possible that you could learn that you have genetic risks for another disease or disability. This may be upsetting and, depending on what you learn, might create a need to make challenging decisions about how to respond.

Although your genomic information is unique to you, you share some genomic similarities with your children, parents, brothers, sisters, and other blood relatives. Therefore, learning your research results could mean something about your family members and might cause you or your

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 




family distress. Before joining the study, it may be beneficial to talk with your family members about whether and how they want you to share your results with them.

# Protections against misuse of genetic information

This study involves genetic testing on samples. Some genetic information can help predict future health problems of you and your family and this information might be of interest to your employers or insurers. The Genetic Information Nondiscrimination Act (GINA) is a federal law that prohibits plans and health insurers from requesting genetic information or using genetic information. It also prohibits employment discrimination based on your health information. However, GINA does not address discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed condition or disease that has a genetic component.

#### WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You might not benefit from being in this study.

However, the potential benefit to you might be shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer.

## Are there any potential benefits to others that might result from the study?

In the future, other people might benefit from this study because of the knowledge gained from this therapeutic intervention.

## WHAT OTHER OPTIONS ARE THERE FOR YOU?

Before you decide whether or not to be in this study, we will discuss other options that are available to you. Instead of being in this study, you could

- choose to be treated with radiation or with drugs already approved by the FDA for your disease
- choose to take part in a different study, if one is available
- choose not to be treated for cancer but you may want to receive comfort care to relieve symptoms.

#### **DISCUSSION OF FINDINGS**

## New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

#### Return of research results

When we are examining your DNA, it is possible that we could identify possible changes in other parts of your DNA that are not related to this research. These are known as "incidental medical findings".

These include:

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




- Changes in genes that are related to diseases other than cancer
- Changes in genes that are not known to cause any disease. These are known as normal variations.
- Changes in genes that are new and of uncertain clinical importance. This means that we do not know if they could cause or contribute to a disease or if they are normal variations.

Since the analyses that we perform in our laboratory are not nearly as sensitive as the tests that are performed in a laboratory that is certified to perform genetic testing, the genetic changes that we find may or may not be valid. Therefore, we do not plan to inform you of all of the genetic results of testing on your tissue and blood that is performed in our research lab. However, in the unlikely event that we discover a finding believed to be clinically important based on medical standards at the time we first analyze your results, we will contact you. This could be many years in the future. We will ask you to provide another sample to verify the findings we have seen in our lab. If the results are verified, you will be re-contacted and offered a referral to a genetic healthcare provider to Discuss the results.

## EARLY WITHDRAWAL FROM THE STUDY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease worsens or comes back during treatment
- if you have side effects from the treatment that your doctor thinks are too severe
- if you become pregnant
- if Minnelide may become unavailable
- if new information shows that another treatment would be better for you
- if you do not follow the study rules
- if the study is stopped for any reason

In this case, you will be informed of the reason therapy is being stopped.

After therapy is stopped we would like to see you for a safety visit 7-30 days after your last dose and before the beginning of a new anti-cancer treatment.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to the Study Sponsor (Center for Cancer Research), Minneamrita Therapeutics or designated representatives.

# STORAGE, SHARING AND FUTURE RESEARCH USING YOUR SPECIMENS AND DATA

#### Will your specimens or data be saved for use in other research studies?

As part of this study, we are obtaining specimens and data from you. We will remove all the identifiers, such as your name, date of birth, address, or medical record number and label your specimens and data with a code so that you cannot easily be identified. However, the code will be linked through a key to information that can identify you. We plan to store and use these

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




specimens and data for studies other than the ones described in this consent form that are going on right now, as well as studies that may be conducted in the future. These studies may provide additional information that will be helpful in understanding ASCP, or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or devices, that may lead to the development of a commercial product by the NIH and/or its research or commercial partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you.

I give permission for my coded specimens and data to be stored and used for future research as described above.

| Yes | No |
|----------|-----------------|
| Initials | <b>Initials</b> |

# Will your specimens or data be shared for use in other research studies?

We may share your coded specimens and data with other researchers. If we do, while we will maintain the code key, we will not share it, so the other researchers will not be able to identify you. They may be doing research in areas that are similar to this study or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or commercial entities.

I give permission for my coded specimens and data to be shared with other researchers and used by these researchers for future research as described above.

| Yes | No |
|----------|----------|
| Initials | Initials |

If you change your mind and do not want us to store and use your specimens and data for future research, you should contact the research team member identified at the top of this document. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your specimens and data. For example, if some research with your specimens and data has already been completed, the information from that research may still be used. Also, for example, if the specimens and data have been shared already with other researchers, it might not be possible to withdraw them.

In addition to the planned use and sharing described above, we might remove all identifiers and codes from your specimens and data and use or share them with other researchers for future research at the NIH or other places. When we or the other researchers access your anonymized data, there will be no way to link the specimens or data back to you. We will not contact you to ask your permission or otherwise inform you before we do this. We might do this even if you answered "no" to the above questions. If we do this, we would not be able to remove your

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




specimens or data to prevent their use in future research studies, even if you asked, because we will not be able to tell which are your specimens or data.

NIH policies require that your clinical and other study data be placed in an internal NIH database that is accessible to other NIH researchers for future research. Usually, these researchers will not have access to any of your identifiers, such as your name, date of birth, address, or medical record number; and your data will be labeled with only a code. We cannot offer you a choice of whether your data to be placed in this database or not. If you do not wish to have your data placed in this database, you should not enroll in this study.

# Will your genomic data be shared outside of this study?

As part of this research study, we will put your genomic data in a large database for broad sharing with the research community. These databases are commonly called data repositories. The information in this database will include but is not limited to genetic information, race and ethnicity, and sex. If your individual data are placed in one of these repositories, they will be labeled with a code and not with your name or other information that could be used to easily identify you, and only qualified researchers will be able to access them. These researchers must receive prior approval from individuals or committees with authority to determine whether these researchers can access the data.

NIH policies require that genomic data be placed in a repository for sharing. Therefore, we cannot offer you a choice of whether your data will be shared. If you do not wish to have your data placed in a repository, you should not enroll in this study.

# How long will your specimens and data be stored by the NIH?

Your specimens and data may be stored by the NIH indefinitely.

# Risks of storage and sharing of specimens and data

When we store your specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity, for example, when appropriate, we remove information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or someone may gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your specimens and data.

#### **PAYMENT**

## Will you receive any type of payment for taking part in this study?

You will not receive any payment for taking part in this study.

#### REIMBURSEMENT

#### Will you receive reimbursement or direct payment by NIH as part of your participation?

On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




If your travel to the NIH Clinical Center (e.g. flight, hotel) is arranged and paid for by the NIH, the agency making the reservations and their representatives will have access to your identifiable information.

#### **COSTS**

## Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

# **CONFLICT OF INTEREST (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

Minneamrita Therapeutics is providing Minnelide for this study to NIH without charge. No NIH employee involved in this study receives any payment or other benefits from Minneamrita Therapeutics.

#### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

## Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor, Center for Cancer Research, or their agent(s)
- Qualified representatives from Minneamrita Therapeutics, the pharmaceutical company who produces Minnelide.

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

#### **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical information that we collect under the authority of the Public Health Service Act. In some cases, the Privacy

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

## POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

## PROBLEMS OR QUESTIONS

| If you have any problems or questions abo | ut this study, or about your rights as a research |
|---|---|
| participant, or about any research-related in | jury, contact the Principal Investigator, Christine |
| Alewine, | . You may also call the NIH Clinical Center |
| Patient Representative at , or the | NIH Office of IRB Operations at , if |
| you have a research-related complaint or conc | em. |

#### CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study




| Signature of Research Participant | Print Name of Researce<br>Participant | ch Date |
|---|---|---|
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| <ul> <li>Witness should sign below if either:</li> <li>1. A short form consent process has been used to enroll a non-English speaking subject or</li> <li>2. An oral presentation of the full consent has been used to enroll a blind or illiterate subject</li> </ul> | | |
| subject or 2. An oral presentation of the | | |
| subject or 2. An oral presentation of the subject | | |
| subject or 2. An oral presentation of the subject Signature of Witness NIH ADMINISTRATIVE SECTIO | Print Name of Witness | Il a blind or illiterate Date |
| subject or 2. An oral presentation of the subject Signature of Witness NIH ADMINISTRATIVE SECTION INTERPRETER: | Print Name of Witness | Date DING THE USE OF |
| subject or 2. An oral presentation of the subject Signature of Witness NIH ADMINISTRATIVE SECTIO AN INTERPRETER: An interpreter, or other individual | Print Name of Witness N TO BE COMPLETED REGAR ual, who speaks English and the pent and served as a witness. The interpretation of the pent and served as a witness. | Date |
| subject or 2. An oral presentation of the subject Signature of Witness NIH ADMINISTRATIVE SECTION INTERPRETER: An interpreter, or other individual language facilitated the administration of informed consent may not also serve as the witness. | Print Name of Witness N TO BE COMPLETED REGAR ual, who speaks English and the pent and served as a witness. The interpretation of the pent and served as a witness. | Date |
| Signature of Witness NIH ADMINISTRATIVE SECTION AN INTERPRETER: An interpreter, or other individual language facilitated the administration of informed conseconsent may not also serve as the witness. | Print Name of Witness N TO BE COMPLETED REGAR ual, who speaks English and the pent and served as a witness. The inness. ual, who speaks English and the pent and served as a witness. | Date Darticipant's preferred investigator obtaining Darticipant's preferred |

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study


